CLINICAL TRIAL: NCT06384547
Title: A Randomized, Controlled, Safety and Tolerability Study of VRDN-001, a Humanized Monoclonal Antibody Directed Against the IGF-1 Receptor, in Participants With Thyroid Eye Disease (TED)
Brief Title: A Randomized, Controlled, Safety and Tolerability Study of VRDN-001 in Participants With Thyroid Eye Disease (TED)
Acronym: STRIVE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Viridian Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VRDN-001-303
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Eye Disease
Keywords: Thyroid Eye Disease; Thyroid-Associated Ophthalmopathy; Dysthyroid Ophthalmopathy; Myopathic Ophthalmopathy; Congestive Ophthalmopathy; Edematous Ophthalmopathy; Infiltrative Ophthalmopathy; Thyroid-Associated Orbitopathy; Graves Disease; Graves Eye Disease; Graves Orbitopathy
MeSH Terms: conditions — Graves Ophthalmopathy; Graves Disease

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, safety and tolerability study of VRDN-001, a humanized monoclonal antibody directed against the IGF-1 receptor, in participants with thyroid eye disease (TED).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- VRDN-001 10 mg/kg (Experimental): 5 infusions of VRDN-001 10 mg/kg
  Interventions: Drug: VRDN-001 10 mg/kg
- 5 infusions of VRDN-001 3 mg/kg (Experimental): 5 infusions of VRDN-001 3 mg/kg
  Interventions: Drug: VRDN-001 3 mg/kg

INTERVENTIONS:
Drug: VRDN-001 10 mg/kg — 5 infusions of VRDN-001 10 mg/kg
  Arms: VRDN-001 10 mg/kg
Drug: VRDN-001 3 mg/kg — 5 infusions of VRDN-001 3 mg/kg
  Arms: 5 infusions of VRDN-001 3 mg/kg

SUMMARY:
The investigational drug, VRDN-001, is a monoclonal antibody that inhibits the activity of a cell surface receptor called insulin-like growth factor-1 receptor (IGF-1R). Inhibition of IGF-1R may help to reduce the inflammation and associated tissue swelling that occurs in patients with thyroid eye disease (TED). The primary objective of this clinical trial is to evaluate the safety and tolerability of VRDN-001 in patients with TED.

DETAILED DESCRIPTION:
A randomized, controlled, safety and tolerability study of VRDN-001, a humanized monoclonal antibody directed against the IGF-1 receptor, in participants with thyroid eye disease (TED).

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of TED with or without proptosis and with any CAS (0 - 7) and in the opinion of the investigator may benefit from treatment
* Must agree to use highly effective contraception method as specified in the protocol
* Female TED participants must have a negative serum pregnancy test
* Not require immediate ophthalmological or orbital surgery in the study eye for any reason

Exclusion Criteria:

* Must not have received prior treatment with another anti-IGF-1R therapy
* Must not have used systemic corticosteroids, or selenium within 2 weeks prior to Day 1
* Must not have received rituximab, tocilizumab or other immunosuppressive agents within 8 weeks prior to Day 1
* Must not have received any other therapy for TED within 8 weeks prior to Day 1
* Must not have received an investigational agent for any condition within 8 weeks prior to the first dose of study medication
* Must not have a pre-existing ophthalmic condition in the study eye that in the opinion of the Investigator would confound interpretation of the study results
* Must not have had previous orbital irradiation or decompression surgery involving excision of fat for TED in the study eye's orbit
* Must not have inflammatory bowel disease
* Must not have abnormal hearing test before first dose. Must also not have a history of ear conditions considered significant by study doctor.
* Must not have received an investigational agent for any condition within 8 weeks prior to Day 1
* Female TED participants must not be pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Event (TEAE) incidence rate | Week 15

SECONDARY OUTCOMES:
Change from baseline in proptosis in the study eye as measured by exophthalmometer | Week 15
Treatment Emergent Adverse Event (TEAE) incidence rate | Week 52

CONTACTS AND LOCATIONS:
Locations (50):
- United States (26):
  - United Medical Research Institute, Inglewood, California
  - Advancing Research International, LLC, Los Angeles, California
  - Stanford Byers Eye Institute, Palo Alto, California
  - Cockerham Eye Consultants, PC, San Diego, California
  - FOMAT Medical Research, Santa Maria, California
  - University of Colorado - Dept of Ophthalmology, Aurora, Colorado
  - Sina Medical Center LLC, Homestead, Florida
  - Med-Care Research Inc., Miami, Florida
  - Edward Jenner Research Group Center LLC, Plantation, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Vision Medical Research Inc., Orland Park, Illinois
  - University Health Diabetes, Endocrinology & Nephrology Center, Kansas City, Kansas
  - KU Medical Center, University of Kansas, Kansas City, Kansas
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Weymouth, Massachusetts
  - Fraser Eye Care Center, Fraser, Michigan
  - Kahana Oculoplastic & Orbital Surgery, Livonia, Michigan
  - University of Minnesota, Department of Ophthalmology and Visual Neurosciences, Minneapolis, Minnesota
  - Advancing Research International, LLC, Las Vegas, Nevada
  - Rutgers- New Jersey Medical School- Newark, Newark, New Jersey
  - New York Eye Ear Infirmary of Mount Sinai, New York, New York
  - Baylor College of Medicine (BCM) - Ophthalmology, Houston, Texas
  - Neuro-Eye Clinical Trials, Houston, Texas
  - Neuro-Ophthalmology of Texas, PLLC, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Australia (2):
  - Sydney Eye Hospital, Sydney
  - North Shore Eye Surgery, Sydney
- France (4):
  - CHU d'Angers, Angers
  - Centre Hospitalier National D'ophtalmologie, Des Quinze Vingts Paris
  - CH Nice, Nice
  - AP-HP - Hôpital de la Pitié Salpétrière, Paris
- Germany (2):
  - Universitätsmedizin Göttingen, Göttingen
  - Johannes Gutenberg-University Medical Center, Mainz
- Poland (5):
  - NZOZ E-Vita, Bialystok
  - Specjalistyczny Osrodek Okulistyczny Oculomedica, Bydgoszcz
  - Santa Familia PTG Lodz, Lódz
  - Panstwowy Instytut Medyczny MSWiA, Warsaw
  - 4 Wojskowy Szpital Kliniczny z Poliklinika SP ZOZ, Wroclaw
- Spain (8):
  - Clinica Bonanova de Cirugia Ocular, Barcelona
  - Hospital Arruzafa, Córdoba
  - Clínica Universidad de Navarra, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Complexo Hospitalario Universitario de Santiago-Hospital Médico-Cirúrxico de Conxo, Santiago de Compostela, A Coruña
  - Hospital Universitario Virgen De La Macarena, Servicio de Oftalmología, Seville
  - Miguel Servet University Hospital, Clinical Trials Unit, Zaragoza
- United Kingdom (3):
  - Northwick Park Hospital, London
  - Western Eye Hospital, Imperial College NHS Trust, London
  - Guy's and St. Thomas NHS Trust, London

IPD SHARING:
Plan to Share IPD: No